CLINICAL TRIAL: NCT06754631
Title: Efficacy and Safety of Continuous Versus Intermittent Nebulization of Salbutamol in Acute Severe Asthma in Children Under 12 Years of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Collaborators: Nishtar Medical University (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHM-1
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Nebulization of Salbutamol (Experimental): The patients received continuous nebulization of salbutamol at a concentration of 0.3 mg/kg/hour for 4 hours, with a minimum of 5 mg/hour and a maximum of 15 mg/hour administered via high-output extended aerosol respiratory therapy (HEART).
  Interventions: Drug: Continuous Nebulization of Salbutamol
- Intermittent Nebulization of Salbutamol (Experimental): The patients were treated with intermittent nebulization of salbutamol at a dose of 0.15 mg/kg/dose, administered through a face mask with an oxygen flow rate of 6-8 L per minute. They received at least 2-3 nebulizations and no more than 7.5 mg/dose every 30 minutes for 4 hours.
  Interventions: Drug: Intermittent Nebulization of Salbutamol

INTERVENTIONS:
Drug: Continuous Nebulization of Salbutamol — Children received continuous nebulization of salbutamol at a concentration of 0.3 mg/kg/hour for 4 hours, with a minimum of 5 mg/hour and a maximum of 15 mg/hour administered via High Output Extended Aerosol Respiratory Therapy (HEART).
  Arms: Continuous Nebulization of Salbutamol
Drug: Intermittent Nebulization of Salbutamol — were treated with intermittent nebulization of salbutamol at a dose of 0.15 mg/kg/dose, administered through a face mask with an oxygen flow rate of 6-8 L per minute. They Children received at least 2-3 nebulizations and no more than 7.5 mg/dose every 30 minutes for 4 hours.
  Arms: Intermittent Nebulization of Salbutamol

SUMMARY:
Asthma affects around 260 million people globally, causing around 0.5 million deaths annually. Pediatric asthma remains a major global public health challenge, significantly affecting the quality of life for many children. Therefore, this study was planned to compare the effects of continuous versus intermittent nebulization of salbutamol in the treatment of acute severe asthma (ASA) in children visiting the emergency department of a tertiary childcare hospital in South Punjab, Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Children of either gender
* Aged 2 to 12 years
* Diagnosed with moderate exacerbation of acute asthma according to British Guidelines on the Management of Asthma, with a clinical asthma score of 8 or more

Exclusion Criteria:

* Children who were prescribed with other first-line therapy, such as adrenaline or 3% NaCl nebulization
* Presented at imminent risk of respiratory arrest
* Congenital heart disease
* Chronic respiratory disease
* Neurological disorders
* Children referred from any other hospital with no data available on emergency treatment

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Discharge | 4 hours
  When patients met the clinical criteria for discharge, which were an asthma score of 5 or less and a saturation level of over 94% on room air.

SECONDARY OUTCOMES:
Hospital stay | 24 hours
  The length of stay in the hospital was calculated from admission to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Arif Zulqarnain, FCPS, Study Director — Children's Hospital and institute of Child Health Multan, Punjab, Pakistan; Muhammad Salman, FCPS, Principal Investigator — Children's Hospital and institute of Child Health Multan, Punjab, Pakistan
Locations (2):
- Pakistan (2):
  - Nishtar Hospital, Multan, Punjab Province
  - The Children's Hospital and The Institute of Child Health, Multan, Punjab Province

IPD SHARING:
Plan to Share IPD: No